CLINICAL TRIAL: NCT01565694
Title: A Phase 3, Open-Label, Baseline-controlled, Multicenter, Sequential Dose Titration Study to Assess the Long-Term Efficacy and Safety, and the Pharmacokinetics of Solifenacin Succinate Suspension in Patients From 5 to Less Than 18 Years of Age With Neurogenic Detrusor Overactivity (NDO)
Brief Title: A Study to Assess the Long Term Effect, Safety and Metabolism of a Solifenacin Liquid Suspension in Participants 5 to 18 Years of Age With Neurogenic Detrusor Overactivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 905-CL-047; 2011-000330-11 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Cognitive Function; Phase 3; Neurogenic Detrusor Overactivity; Pharmacokinetics; Ocular Accommodation; Urodynamics
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Solifenacin succinate (Experimental): Participants aged 5 years to < 18 years received solifenacin orally once a day, with sequential titrated doses for 12 weeks to identify the optimal dose during the dose-titration period. The initial dose was pediatric equivalent dose (PED) 5 mg.
  After completing the dose titration period participants entered the fixed-dose period during which solifenacin was taken orally once a day for 40 weeks or until the end of study visit (Week 52).
  Interventions: Drug: Solifenacin succinate

INTERVENTIONS:
Drug: Solifenacin succinate — Oral suspension administered once a day via syringe.
  Other Names: YM905

SUMMARY:
The purpose of this study was to investigate a medicine for the treatment of symptoms and complications of neurogenic detrusor overactivity (NDO) in children and adolescents.

DETAILED DESCRIPTION:
The NDO often occurs in patients with spina bifida or other spinal cord damage where the bladder muscle contracts more than normal during filling. These patients often have an inability to void, so that catheterization is required to empty the bladder.

The medicine being tested in this study is called solifenacin succinate. Solifenacin tablets are given to adults for the treatment of overactive bladder. A new liquid suspension has been developed to treat children and adolescents in this and other studies.

The efficacy and safety of the solifenacin suspension was investigated. The take-up and length of time that the solifenacin suspension stays in the body was also investigated during this study. Effectiveness was measured by urodynamics (the filling and emptying of the bladder) and the urine volumes during catheterization together with the diary responses relating to the number of incontinence episodes or incontinence free days.

Safety assessments included analysis of the blood and urine, review of the electrocardiogram (ECG), ultrasound of the kidney, simple memory and understanding tests (cognitive function) and the ability to see near and far objects (visual accommodation).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of NDO, confirmed by urodynamics
* Practicing clean intermittent catheterization (CIC)
* Currently on treatment with an antimuscarinic drug

Exclusion Criteria:

* Known genitourinary condition (other than NDO) that may cause incontinence
* Bladder augmentation surgery
* Current Faecal impaction
* Electro-stimulation therapy within 2 weeks prior to screening and at any time during the study
* Subjects with the following gastro-intestinal problems: partial or complete obstruction, decreased motility like paralytic ileus, subjects at risk of gastric retention
* Reflux grade 3 or 4
* Current urinary tract infection (UTI)
* Subject has severe renal impairment (glomerular filtration rate < 30 ml/min)
* Subject has severe hepatic impairment (Child-Pugh score > 9).
* Subject has received intra-vesical botulinum toxin within 9 months prior to screening

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (21):
- United States (2):
  - Site US1008, Tarrytown, New York
  - Site US1010, Cincinnati, Ohio
- Site BE3201, Ghent, Belgium
- Brazil (5):
  - Site BR5505, São José do Rio Preto, São Paulo
  - Site BR5507, Campinas
  - Site BR5504, Campinas
  - Site BR5506, Curitiba
  - Site BR5503, Porto Alegre
- Site DK4501, Aarhus, Denmark
- Site HU3602, Miskolc, Hungary
- Mexico (2):
  - Site MX5203, León
  - Site MX5205, Mexico City
- Philippines (2):
  - Site PH6301, Manila
  - Site PH6302, Quezon City
- Poland (3):
  - Site PL4803, Gdansk
  - Site PL4805, Gdansk
  - Site PL4801, Warsaw
- South Korea (2):
  - Site KR8207, Seoul
  - Site KR8201, Seoul
- Turkey (Türkiye) (2):
  - Site TR9003, Ankara
  - Site TR9002, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Tannenbaum S, den Adel M, Krauwinkel W, Meijer J, Hollestein-Havelaar A, Verheggen F, Newgreen D. Pharmacokinetics of solifenacin in pediatric populations with overactive bladder or neurogenic detrusor overactivity. Pharmacol Res Perspect. 2020 Dec;8(6):e00684. doi: 10.1002/prp2.684. PMID 33231929
- [Derived] Franco I, Hoebeke P, Baka-Ostrowska M, Bolong D, Davies LN, Dahler E, Snijder R, Stroosma O, Verheggen F, Newgreen D, Bosman B, Vande Walle J. Long-term efficacy and safety of solifenacin in pediatric patients aged 6 months to 18 years with neurogenic detrusor overactivity: results from two phase 3 prospective open-label studies. J Pediatr Urol. 2020 Apr;16(2):180.e1-180.e8. doi: 10.1016/j.jpurol.2019.12.012. Epub 2019 Dec 27. PMID 32007426
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of male and female participants with neurogenic detrusor overactivity (NDO) aged 5 years to < 18 years old.
Pre-assignment Details: After screening and a 14-day washout period, participants were treated with sequential doses of solifenacin oral suspension for 12 weeks (titration period) to determine each participant's optimal dose, after which a fixed dose of solifenacin oral suspension was given for at least 40 weeks (fixed dose assessment period).
Groups:
- Solifenacin Succinate: Participants aged 5 years to < 18 years, received solifenacin orally once a day, with sequential titrated doses for 12 weeks, to identify optimal dose during dose-titration period. After completing dose titration period, participants entered fixed-dose period during which solifenacin was received orally once a day for 40 weeks or until the end of study visit (Week 52).
Period: Dose-Titration Period
Arm/Group | Solifenacin Succinate
Started | 76
Completed | 62
Not Completed | 14
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 10
Period: Fixed-Dose Assessment Period
Arm/Group | Solifenacin Succinate
Started | 62
Completed | 58
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who had a baseline and 1 post baseline measurement for the primary endpoint (MCC) and have received at least 1 dose of study drug.
Groups:
- Solifenacin Succinate: Participants aged 5 years to < 18 years, received solifenacin orally once a day, with sequential titrated doses for 12 weeks to identify optimal dose during the dose-titration period. After the dose titration period participants entered the fixed-dose period and received a fixed dose of solifenacin once a day orally for 40 weeks or until the end of study visit (Week 52).
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.8 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 37
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 65
Race [Count of Participants; unit: Participants]
  White | 45
  Black/African American | 2
  Asian | 23
  American Indian/Alaskan Native | 1
  Other | 5
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 38.1 (15.5)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 138 (16.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m^2)] | 19.2 (4.69)
Duration of Neurogenic Detrusor Overactivity (NDO) Disease [Median (Full Range); unit: Years] | 8.24 [0.4 to 16.2]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Maximum Cystometric Capacity (MCC)
Description: During urodynamic assessments, the bladder was filled until voiding/leakage begins, or until it was stopped because either the participant experiences pain or discomfort or 135% of expected bladder capacity for age has been reached. MCC is the maximum bladder capacity reached during filling cystometry before either leakage or pain/discomfort was observed.
Time Frame: Baseline and Week 24
Population: The full analysis set (FAS) consisted of all participants who had a baseline and 1 post baseline measurement for the primary endpoint (MCC) and have received at least 1 dose of study drug. Last observation carried forward (LOCF) was utilized.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Solifenacin Succinate: Participants aged 5 years to < 18 years, received solifenacin orally once a day, with sequential titrated doses for 12 weeks, to identify optimal dose during the dose-titration period. After completing dose titration period, participants entered the fixed-dose period during which solifenacin was received orally once a day for 40 weeks or until the end of study visit (Week 52).
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 55
mL
  Change from Baseline Week 24: number analyzed (Participants) | 49
  Change from Baseline Week 24 | 57.2 (107.7)
  Change from Baseline Week 24 (LOCF) | 59.3 (107.5)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Change From Baseline to Last Possible Titration Step in Maximum Cystometric Capacity
Description: During urodynamic assessments, the bladder was filled until voiding/leakage begins, or until it was stopped because either the participant experiences pain or discomfort or 135% of expected bladder capacity for age has been reached. MCC is the maximum bladder capacity reached during filling cystometry before either leakage or pain/discomfort was observed. Based on study requirements, the last possible titration step was Week 9 for participants enrolled under versions 1.0 and 1.1 and Week 12 under later versions.
Time Frame: Baseline, Week 9 or Week 12
Population: The full analysis set (FAS) consisted of all participants who had a baseline and 1 post baseline measurement for the primary endpoint (MCC) and have received at least 1 dose of study drug. The number of participant analyzed represents participants with a non-missing change from baseline to last possible titration step.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 50
mL | 57.4 (105.5)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Test type: Other — P-Value was obtained from a 2-sided one sample t-test, testing the null hypothesis that Change from Baseline=0; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Bladder Compliance
Description: Bladder compliance gives an indication of the elasticity of the bladder wall and was calculated by dividing the change in volume by the change in detrusor pressure during the filling of the bladder.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
mL/cmH2O
  Change from Baseline Week 24: number analyzed (Participants) | 50
  Change from Baseline Week 24 | 9.1 (28.6)
  Change from Baseline Week 24 (LOCF): number analyzed (Participants) | 53
  Change from Baseline Week 24 (LOCF) | 8.8 (27.8)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.029, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.026, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Bladder Volume (mL) Until First Detrusor Contraction > 15 cmH2O as a Percentage of Expected Bladder Capacity (EBC)
Description: Change from baseline in the bladder volume was calculated using urodyanamic assessments. During urodynamic assessments, the bladder is filled until voiding/leakage begins, or until it is stopped because either the subject experiences pain or discomfort or 135% of expected bladder capacity for age has been reached. If no detrusor contraction of at least 15 cmH2O occurs, the bladder volume was imputed with MCC.
Time Frame: Baseline and Week 24
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Percentage of EBC
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 50
Percentage of EBC | 23.10 [-117.2 to 114.7]
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — From a Wilcoxon Signed Rank testing the null hypothesis is that the Median at Week 24 is equal to Baseline Median; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline in Bladder Volume at 30 cmH2O Detrusor Pressure
Description: Bladder volumes at 30 cm H2O detrusor pressure was calculated using the urodynamic assessments. During urodynamic assessments, the bladder is filled until voiding/leakage begins, or until it is stopped because either the participants experiences pain or discomfort or 135% of expected bladder capacity for age has been reached.
Time Frame: Baseline and Week 24
Population: The full analysis set (FAS) consisted of all participants who had a baseline and 1 post baseline measurement for the primary endpoint (MCC) and have received at least 1 dose of study drug. Last observation carried forward (LOCF) was utilized. Only participants who reached 30 cmH20 detrusor pressure were included in the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 25
mL
  Change from Baseline Week 24: number analyzed (Participants) | 17
  Change from Baseline Week 24 | 61.8 (80.6)
  Change from Baseline Week 24 (LOCF): number analyzed (Participants) | 21
  Change from Baseline Week 24 (LOCF) | 71.9 (88.3)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 in bladder volume at 30 cmH20; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.006, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF in bladder volume at 30 cmH20; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.001, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Bladder Volume at 40 cmH2O Detrusor Pressure
Description: Bladder volumes at 40 cm H2O detrusor pressure were calculated using urodynamic assessments. During urodynamic assessments, the bladder is filled until voiding/leakage begins, or until it is stopped because either the subject experiences pain or discomfort or 135% of expected bladder capacity for age has been reached.
Time Frame: Baseline and Week 24
Population: The full analysis set (FAS) consisted of all participants who had a baseline and 1 post baseline measurement for the primary endpoint (MCC) and have received at least 1 dose of study drug. Last observation carried forward (LOCF) was utilized. Only participants who reached 40 cmH20 detrusor pressure were included in the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 18
mL
  Change from Baseline Week 24: number analyzed (Participants) | 10
  Change from Baseline Week 24 | 67.0 (44.3)
  Change from Baseline Week 24 (LOCF): number analyzed (Participants) | 12
  Change from Baseline Week 24 (LOCF) | 54.4 (52.9)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to week 24 in bladder volume at 40 cmH20; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to week 24 LOCF in bladder volume at 40 cmH20; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.004, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Number of Overactive Detrusor Contractions (> 15 cmH2O) Until End of Bladder Filling
Description: Change from baseline in number of overactive detrusor contractions until end of bladder filling was measured by urodynamic testing. If leakage occurred, the "Detrusor pressure at leakage" was recorded otherwise the volume of fluid instilled into the bladder was recorded.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Detrusor Contractions
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
Detrusor Contractions
  Change from Baseline Week 24: number analyzed (Participants) | 50
  Change from Baseline Week 24 | -2.3 (5.1)
  Change from Baseline Week 24 (LOCF) | -1.8 (6.0)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.003, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.028, t-test, 2 sided

8. Secondary Outcome: Change From Baseline in Detrusor Pressure at the End of Bladder Filling
Description: The bladder was filled until voiding/leakage began or until it was stopped because either the participant experiences pain or discomfort or 135% of expected bladder capacity for age has been reached. Pressure was recorded for an extra 5 minutes after leakage began or the end of bladder-filling, whichever is sooner.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 51
cmH2O
  Change from Baseline Week 24: number analyzed (Participants) | 46
  Change from Baseline Week 24 | -9.2 (33.6)
  Change from Baseline Week 24 (LOCF) | -8.2 (32.2)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.068, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.075, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Average Catheterized Volume Per Catheterization
Description: The average catheterized volume per catheterization was calculated using all available (non-zero) catheterized volumes recorded over both of the 2 measuring days in the diary, whether or not these 2 days are concurrent.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
mL
  Change from Baseline Week 24: number analyzed (Participants) | 51
  Change from Baseline Week 24 | 46.23 (48.32)
  Change from Baseline Week 24 (LOCF) | 48.86 (50.98)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Change From Baseline in Maximum Catheterized Volume
Description: The maximum catheterized volume per day was calculated using all available (non-zero) catheterized volumes recorded for the 2 measuring days in the diary, whether or not these 2 days were concurrent. The maximum value was calculated separately for each measuring day and the mean of these two values was used.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
mL
  Change from Baseline Week 24: number analyzed (Participants) | 51
  Change from Baseline Week 24 | 67.45 (88.07)
  Change from Baseline Week 24 (LOCF) | 69.63 (88.84)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Average First Morning Catheterized Volume
Description: The average first morning catheterized volume was calculated as the average of the available first morning catheterized volumes recorded for the 2 measuring days in the diary, whether or not these 2 days are concurrent.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
mL
  Change from Baseline Week 24: number analyzed (Participants) | 51
  Change from Baseline Week 24 | 43.24 (72.78)
  Change from Baseline Week 24 (LOCF) | 44.21 (73.40)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Mean Number of Incontinence Episodes Per 24 Hours
Description: The mean of the number of incontinence episodes per 24h was calculated as the mean over the valid diary days in the 7-day diary.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
Incontinence Episodes
  Change from Baseline Week 24: number analyzed (Participants) | 51
  Change from Baseline Week 24 | -1.60 (2.04)
  Change from Baseline Week 24 (LOCF) | -1.62 (2.04)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Number of Dry (Incontinence-Free) Days Per 7 Days
Description: The number of incontinence-free days was calculated from the 7-day micturition diary.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
Days
  Change from Baseline Week 24: number analyzed (Participants) | 51
  Change from Baseline Week 24 | 1.06 (2.83)
  Change from Baseline Week 24 (LOCF) | 1.19 (2.86)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.010, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.004, t-test, 2 sided

14. Secondary Outcome: Change From Baseline in Number of Dry (Incontinence-Free) Nights Per 7 Days
Description: The number of incontinence-free nights was calculated from the 7-day micturition diary.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nights
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 54
Nights
  Change from Baseline Week 24: number analyzed (Participants) | 51
  Change from Baseline Week 24 | 1.60 (3.08)
  Change from Baseline Week 24 (LOCF) | 1.64 (3.06)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p < 0.001, t-test, 2 sided

15. Secondary Outcome: Change From Baseline in Quality of Life [QoL] (PinQ Questionnaire Score)
Description: Pediatric Incontinence Questionnaire (PinQ) is a 20-item questionnaire addressing quality of life for participants with bladder disorders. Each question was answered on a scale from 0 (no, never) to 4 (all the time). The total score ranged from 0 to 80, with higher scores indicated more impact on the quality of life.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 55
Units on a Scale
  Change from Baseline Week 24: number analyzed (Participants) | 53
  Change from Baseline Week 24 | -0.7 (8.3)
  Change from Baseline Week 24 (LOCF): number analyzed (Participants) | 51
  Change from Baseline Week 24 (LOCF) | -0.7 (8.3)
Statistical Analysis 1: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.568, t-test, 2 sided
Statistical Analysis 2: Comparison: Solifenacin Succinate; Analysis of change from baseline to Week 24 LOCF; Test type: Other — P-Value was calculated from a 2-sided one sample t-test, testing the null hypothesis that change from baseline = 0; p = 0.573, t-test, 2 sided

16. Secondary Outcome: Number of Participants With Adverse Events
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event observed after starting administration of the first dose of study medication on Day 1. All adverse events collected within 7 days after taking the last dose of study drug were counted as a TEAE.
Time Frame: Baseline to End of Study Visit (Week 52)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Solifenacin Succinate
Number analyzed (Participants) | 76
Participants
  TEAEs | 51
  Drug related TEAE | 15
  Deaths | 0
  Serious TEAEs | 7
  Drug related Serious TEAEs | 0
  TEAEs Leading to Discontinuation | 4
  Drug related TEAEs Leading to Discontinuation | 3

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to the last dose of study drug (up to week 52).
Arm/Group | Solifenacin Succinate
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 7/76
Other Adverse Events (participants affected / at risk) | 42/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solifenacin Succinate (N=76)
Tachycardia (Cardiac disorders) | 1 (1)
Megacolon (Gastrointestinal disorders) | 1 (2)
Dengue fever (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Tethered cord syndrome (Nervous system disorders) | 1 (1)
Spinal cord operation (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solifenacin Succinate (N=76)
Constipation (Gastrointestinal disorders) | 6 (10)
Escherichia urinary tract infection (Infections and infestations) | 6 (7)
Nasopharyngitis (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (6)
Urinary tract infection (Infections and infestations) | 12 (12)
Urinary tract infection bacterial (Infections and infestations) | 14 (17)
Electrocardiogram QT prolonged (Investigations) | 4 (4)
Headache (Nervous system disorders) | 4 (4)
Bladder pain (Renal and urinary disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor at least 1 month prior to the submission of any such information to an editorial board or scientific review committee. This allows the Sponsor to protect proprietary information and to provide comments based on information from other studies that may not yet be available to the investigator.